CLINICAL TRIAL: NCT04772846
Title: Adjuvant Chloroquine to the Conventional Treatment for Glioblastoma.
Brief Title: Chloroquine for Glioblastoma.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Egyptian Medical Syndicate (Other)
Responsible Party: Principal Investigator, Mohammed A. Azab, Department of Neurosurgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CQGBM
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Tablets

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroquine group (Experimental)
  Interventions: Drug: Oral tablet
- Placebo drug group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral tablet — Oral 250mg chloroquine tablets
  Arms: Chloroquine group
Drug: Placebo — Oral placebo tablets
  Arms: Placebo drug group

SUMMARY:
Adjuvant chloroquine to the conventional treatment for glioblastoma; A randomized, single-blind, placebo-controlled, phase I/II trial.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed glioblastoma Adequate hematologic, hepatic, and renal function Karnofsky performance status score ≥ 70% Life expectancy ≥ six weeks

Exclusion Criteria:

Abnormal severe un-controlled medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Survival duration after surgery | Three years

SECONDARY OUTCOMES:
End-point evaluation, survival at three years | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Private clinics, Cairo, Egypt